CLINICAL TRIAL: NCT02223975
Title: Evaluation of the Role of Vibrational Spectroscopy in the Assessment of Vulval Disease
Acronym: Vulval VS
Status: Suspended | Type: Observational
Why Stopped: Study suspended pending further funding
Sponsor: Gloucestershire Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Jonathan Frost, Clinical Research Fellow, Gloucestershire Hospitals NHS Foundation Trust
Other Study IDs: 14/040/GHT
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Normal Vulval Skin; Lichen Sclerosus; High Grade Dysplasia - Usual Type ('VIN 2-3'); High Grade Dysplasia - Differentiated Type ('VIN 2-3'); Squamous Cell Carcinoma; Epithelial Hyperplasia Without Atypia; Atypia Not Otherwise Specified/ Low Grade Dysplasia ('VIN 1'); Pagets Disease of the Vulva
Keywords: Spectrum Analysis, vibrational; Spectrum Analysis, infrared; Spectrum Analysis, Raman; Spectrum Analysis; Fourier transform infrared spectroscopy; Raman probe; Optical; Diagnosis; Cancer; Multivariate analysis; Vulval Intraepithelial Neoplasia; Vulvar Neoplasm; Vulva; Vulvar Diseases
MeSH Terms: conditions — Lichen Sclerosus et Atrophicus; Carcinoma, Squamous Cell; Disease; Neoplasms; Vulvar Neoplasms; Vulvar Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Histological sections of vulval and lymph node tissue.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vulval Disease: Patients who have undergone vulval skin biopsy or surgery for a vulval condition within Gloucestershire Hospitals NHS Foundation Trust.

SUMMARY:
Can vibrational spectroscopy be used to accurately assess vulval skin conditions? Vulval skin disorders are common and the diagnosis of these conditions can be difficult. Reliable discrimination between benign vulval skin conditions, precancerous conditions or vulval cancer often requires tissue biopsies. In addition the monitoring of patients with vulval disease at risk cancerous change is currently limited to visual assessment often supplemented by multiple invasive tissue biopsies. There are currently no established non invasive tests available for the diagnosis of vulval skin diseases.

The vibrational spectroscopic techniques of Raman spectroscopy and Fourier transform infrared spectroscopy are non invasive diagnostic tools that use the interaction of light within tissues to identify the chemical composition of different tissues. The use of these tools may reduce the need for invasive biopsies to diagnose and monitor women with vulval skin disease.

The aim of this project is to explore the use of vibrational spectroscopic techniques in the diagnosis of vulval skin disease. This will be achieved by performing vibrational spectroscopy on samples of tissue previously taken from women with vulval skin disease treated at Gloucestershire Hospitals NHS Foundation Trust. The results of the spectroscopy will be compared with the routine tests and the accuracy of spectroscopy determined.

DETAILED DESCRIPTION:
Design Ex vivo vibrational spectroscopic analysis of existing stored vulval and lymph node tissue samples collected from patients who have undergone treatment for vulval disease. Vibrational spectra are to be correlated with consensus histopathology and multivariate analysis to be used to evaluate the classification accuracy of vibrational spectroscopy ex vivo.

Aims

1. To establish vibrational spectral signal characteristics across a range of known vulval skin conditions.
2. To evaluate the ability of vibrational spectroscopic techniques to differentiate different vulval skin conditions.
3. To evaluate the ability of vibrational spectroscopy to detect diseased lymph nodes in women who have undergone surgery for vulval cancer.
4. To further the understanding of biochemical changes in a range of known vulval skin conditions.

ELIGIBILITY:
Inclusion Criteria:

* Vulval skin tissue stored after routine histopathological analysis from women treated or investigated for a vulval skin condition.
* Inguinofemoral lymph nodes stored after routine histopathological analysis from women treated for vulval cancer.

Exclusion Criteria:

* Tissue specimens inadequate for analysis.

Ages: 16 Years to 120 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have undergone vulval skin biopsy or surgery for a vulval condition within Gloucestershire Hospitals NHS Foundation Trust.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-08; Primary Completion 2018-08-01 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of vibrational spectroscopic techniques for differentiating key vulval tissue types | 2 years
  * Normal vulval skin
  * Lichen Sclerosus
  * High grade dysplasia - Usual type ('Vulval Intraepithelial Neoplasia 2-3')
  * High grade dysplasia - Differentiated type ('Vulval Intraepithelial Neoplasia 2-3')
  * Squamous cell carcinoma
Diagnostic performance of vibrational spectroscopic techniques for differentiating between normal and diseased lymph nodes in vulval carcinoma. | 2 years
  Diagnostic performance of vibrational spectroscopic techniques for differentiating between normal and diseased lymph nodes in vulval carcinoma.

SECONDARY OUTCOMES:
Diagnostic performance of vibrational spectroscopic techniques for differentiating other vulval tissue types | 2 years
  * Epithelial hyperplasia without atypia
  * Atypia not otherwise specified/ Low grade dysplasia ('VIN 1')
  * Pagets disease of the vulva

CONTACTS AND LOCATIONS:
Locations (1):
- Gloucestershire Hospitals NHS Foundation Trust, Gloucester, Gloucestershire, United Kingdom